CLINICAL TRIAL: NCT01420341
Title: A Comparison Between 12 vs. 20 Weeks of Co-trimoxazole as Maintenance Therapy for Melioidosis
Brief Title: Co-trimoxazole as Maintenance Therapy for Melioidosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Siriluck Anunnatsiri, MD, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE541074; project number 542040 (Other Grant/Funding Number: Khon Kaen University); 106698/B/14/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Melioidosis
Keywords: Melioidosis; Co-trimoxazole; Relapse
MeSH Terms: conditions — Melioidosis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-trimoxazole 12 (Active Comparator): Receive treatment with co-trimoxazole for 12 weeks.
  Interventions: Drug: Co-trimoxazole 12
- Co-trimoxazole 20 (Experimental): Receive treatment with co-trimoxazole for 20 weeks.
  Interventions: Drug: Co-trimoxazole 20

INTERVENTIONS:
Drug: Co-trimoxazole 12 — Receive treatment with co-trimoxazole for 12 weeks.
  Arms: Co-trimoxazole 12
Drug: Co-trimoxazole 20 — Receive treatment with co-trimoxazole for 20 weeks.
  Arms: Co-trimoxazole 20

SUMMARY:
This is a randomised, open-labelled, controlled trial to compare the efficacy and effectiveness on relapse-free rate of 12-week versus 20-week oral eradication treatment of melioidosis. The study population includes 800 patients with culture-confirmed melioidosis whom 12 weeks of oral eradication therapy have been completed with or without intravenous intensive antibiotics. Patients will be randomised to either stop the eradication treatment or continue current oral treatment for 8 more weeks. The study aim to optimise the regimen used to treat melioidosis for better compliance and reducing unnecessary use of antibiotics.

DETAILED DESCRIPTION:
Planed interim analysis will be conducted when the patient enrollment reaches 600 cases for evaluating safety and futility of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 15 years
2. Culture-confirmed melioidosis
3. Currently on oral co-trimoxazole for 12(+2) weeks without any clinical evidence of active melioidosis
4. High likelihood of completing at least 6 months follow up
5. Willingness to participate in the study and written, informed consent obtained from the patient

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Contraindications to TMP-SMX: G6PD, severe adverse reactions grade 3-4 occurring during first 12 weeks of treatment
3. Relapse melioidosis with at least 2 year symptom free period from last episode

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2011-08; Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
1-year non relapse rate | 1 year
  This is defined as clinical features of melioidosis after initial improvement, in association with cultures from any site positive for Burkhoderia pseudomallei. This can be any time point during or after stopping antibiotic treatment.

SECONDARY OUTCOMES:
Clinical Recurrence | 1 year
  Recurrent clinical features of melioidosis treated as such but not confirmed by positive culture.
Treatment failure | 9 weeks
  Clinical decision to change treatment according to inadequate response to therapy.
Mortality | 1 year
Adverse Drug Reactions | 9 weeks
  Adverse events that are caused by the drug including drug allergy.
Drug compliance | 12 or 20 weeks
  This will be done by interviewing and pill counting.

CONTACTS AND LOCATIONS:
Overall Officials: Siriluck Anunnatsiri, MD, Principal Investigator — Khon Kaen Univerisity
Locations (1):
- Khon Kaen Univerisity, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anunnatsiri S, Chaowagul W, Teparrukkul P, Chetchotisakd P, Tanwisaid K, Khemla S, Narenpitak S, Pattarapongsin M, Kongsawasd W, Pisuttimarn P, Thipmontree W, Mootsikapun P, Chaisuksant S, Chierakul W, Day NPJ, Limmathurotsakul D. A Comparison Between 12 Versus 20 Weeks of Trimethoprim-sulfamethoxazole as Oral Eradication Treatment for Melioidosis: An Open-label, Pragmatic, Multicenter, Non-inferiority, Randomized Controlled Trial. Clin Infect Dis. 2021 Dec 6;73(11):e3627-e3633. doi: 10.1093/cid/ciaa1084. PMID 32725199